CLINICAL TRIAL: NCT04458233
Title: FNA Guided Ultrasonography Needle Technique Axial Vs Lateral Approach Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 0006-20
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long axis (Active Comparator)
  Interventions: Procedure: long axis FNA method
- short axis (Active Comparator)
  Interventions: Procedure: long axis FNA method

INTERVENTIONS:
Procedure: long axis FNA method — ). A "long-axis" view (i.e., a longitudinal image of the needle) is obtained by placing the US probe in a parallel position relative to the course of the needle. Short-axis and long-axis views can be used for both US assistance and guidance of FNA procedure. Correspondingly, approaching the nodule with the needle from the lateral or frontal aspect results in either a long axis or short axis view of the needle on the US screen
  Other Names: short axis FNA method

SUMMARY:
Ultrasound-guided fine needle aspiration cytology (FNAC) has been proven to be an accurate and efficient tool in thyroid nodule evaluation. Thyroid nodule aspiration is performed by the use of either two techniques; the short axis approach by which only the tip of the needle is observed, or the long axis approach by which the entire needle is observed. Controversial remains of which approach produces better diagnostic adequacy and less non-diagnostic (Bethesda category I) results.

DETAILED DESCRIPTION:
200 patients presenting electively for thyroid FNA will recruited. Patients will be randomly assigned to two groups: short axis or long axis FNA. FNA will be performed by a single physician at the Ziv medical center ENT clinics.

patient group randomization will be performed according to a random number sequence generated by the SPSS system. Randomization will be performed on admission prior to the procedure.

FNAC sample diagnosis will be performed according to the regular protocol. Laboratory personnel will be blinded to the sample group.

sample results will be compared and analyzed. A P value of less than 0.05 will be regarded as significant.

ELIGIBILITY:
Inclusion Criteria:

* suspected thyroid nodule requiring diagnostic FNA,

Exclusion Criteria:

* under or above age limit, no informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
amount of FNAC non diagnostic Bethesda 1 results | 1 year
  The exact preferred technique for performing Ultrasound Guided FNA is unclear. The correct positioning of the US probe and or the FNA needle could have a marked effect on the diagnostic results of the biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: No
no individual data to be shared